CLINICAL TRIAL: NCT06837974
Title: Construction and Application of an AI Model for Guided TIPS Surgical Puncture: a Prospective Multicenter Randomized Controlled Trial
Brief Title: AI-guided TIPS Procedure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GPS-TIPS001
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Portal Hypertension Related to Cirrhosis
Keywords: TIPS; AI; Efficacy; Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI guided TIPS (Experimental): TIPS procedure will be conducted under the guidance of AI model
  Interventions: Other: AI guided TIPS
- Artificially blinded TIPS (Placebo Comparator): TIPS will be conducted based on the experience of operators.
  Interventions: Other: Artificially blinded TIPS

INTERVENTIONS:
Other: AI guided TIPS — The TIPS procedure will be conducted under the guidance of AI model which was constructed based on the pre-operation enhanced CT images and intra-operation DSA images.
  Arms: AI guided TIPS
Other: Artificially blinded TIPS — The TIPS procedure will be conducted based on the experience of operators.
  Arms: Artificially blinded TIPS

SUMMARY:
The goal of this clinical trial is to learn if transjugular intrahepatic portosystemic shunt (TIPS)-guided AI model can guide TIPS procedure in adults better than conventional TIPS procedure (artificially blinded TIPS). TIPS surgical outcomes and intraoperative and postoperative complications will also be observed. The main questions it aims to answer are:

* Does the AI model lower the number of punctures, radiation dose, and complications of participants undergo TIPS?
* Does the AI model improve the efficacy of TIPS for participants?

Participants will:

* Take the TIPS by the guidance of the AI model or conventional manually blinded penetration (placebo)
* The number of punctures, the success rate of the procedure, the radiation dose, intraoperative complications and postoperative complications within 3 months will be recorded
* Intraoperative portal pressure gradient drop values, symptoms of ascites and rebleeding within 3 months after TIPS will be reported

ELIGIBILITY:
Inclusion Criteria:

* Participants who require transjugular intrahepatic portosystemic shunt (TIPS) and meet the clinical indications for the procedure.
* Participants whose physical condition is suitable for TIPS.

Exclusion Criteria:

* Participants with a history of allergy or serious adverse reactions to iodine contrast media or other related drugs.
* Participants are pregnant or breastfeeding.
* Participants are unwilling or unable to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of punctures | From the beginning to the end of the TIPS procedure.
  The number of punctures is defined as the number of punctures to the liver during the establishment of the puncture channel during the TIPS procedure.

SECONDARY OUTCOMES:
Radiation dose | From the beginning to the end of the TIPS procedure.
  Radiation dose from the TIPS procedure.
Surgical success rate | From the beginning to the end of the TIPS procedure.
  Procedural success was defined as the success of placing a stent and reducing the portal pressure gradient during the TIPS procedure
Complications | From enrollment to the end of the TIPS procedure at 3 months.
  Complications are defined as bleeding, infection, and other complications due to puncture.

OTHER OUTCOMES:
Portal pressure gradient | From the beginning to the end of the TIPS procedure.
  The hepatic venous pressure gradient (HVPG) is an indirect method of assessing the portal pressure gradient by determining the difference between wedged hepatic venous pressure (WHVP) and free hepatic venous pressure (FHVP). pressure (FHVP), which reflects the pressure difference between the portal vein and the intra-abdominal vena cava.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Wuhan Union Hospital, Wuhan, Hubei
  - Wuhan Union Jinyinhu Hospital, Wuhan, Hubei
  - Wuhan Union West Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No